CLINICAL TRIAL: NCT00943449
Title: A Proof-of-concept Phase II Study to Evaluate Efficacy, Safety and Pharmacokinetics of 4SC-201 and the Treatment Combination of Sorafenib Plus 4SC-201 in Patients With Hepatocellular Carcinoma Exhibiting Progressive Disease Under Sorafenib Treatment
Brief Title: 4SC-201 (Resminostat) and Sorafenib in Advanced Hepatocellular Carcinoma
Acronym: Shelter
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-201-1-2009
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; HDAC; 4SC-201; Phase II; Resminostat
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

ARMS (2):
- 4SC-201 (Experimental)
  Interventions: Drug: 4SC-201
- 4SC-201 + Sorafenib (Experimental)
  Interventions: Drug: 4SC-201; Drug: Sorafenib

INTERVENTIONS:
Drug: 4SC-201 — oral administration
Drug: Sorafenib — oral administration
  Arms: 4SC-201 + Sorafenib

SUMMARY:
The purpose of the study is to determine whether 4SC-201 alone or in combination with Sorafenib is effective and safe in the treatment of hepatocellular carcinoma in patients refractory to Sorafenib monotherapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Advanced stage hepatocellular carcinoma
* Patients exhibiting progressive disease under Sorafenib treatment
* Child-Pugh class A and B. Only patients with Child-Pugh index class B of not more than 7 will be included
* ECOG performance status 0, 1 or 2
* Precedent first-line treatment with Sorafenib minimum continuous dosing of 400 mg per day for at least 8 weeks

Main Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1) - any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring hemo- or peritoneal dialysis
* Known central nervous system (CNS) tumors including symptomatic brain metastasis
* Child-Pugh index class B in combination with more than slight ascites or hepatic encephalopathy > Grade I
* Pregnant or breastfeeding women
* Sorafenib intolerance
* Major surgery within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival Rate (PFSR) of repeated oral doses of 4SC-201 and of the treatment combination of Sorafenib plus 4SC-201 | 12 weeks

SECONDARY OUTCOMES:
To establish the MTD of 4SC-201 in combination with Sorafenib | 12 weeks
To investigate the safety and tolerability of repeated oral doses of 4SC-201 and of the treatment combination of ascending repeated oral doses of 4SC-201 and Sorafenib | 12 weeks
To investigate biomarkers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bitzer, Prof. MD, Principal Investigator — Medizinische Universitäts-Klinik Tübingen
Locations (15):
- Germany (8):
  - ONKOPLUS Beratung und Hilfe für Menschen mit Krebs, Berlin
  - Universitätsklinikum Essen (Innere Klinik/Tumorforschung und Zentrum für Innere Medizin), Essen
  - Medizinische Fakultät der Martin-Luther-Universität Halle-Wittenberg (Klinik und Poliklinik für Innere Medizin I), Halle
  - Universitätsklinikum Hamburg-Eppendorf (I. Medizinische Klinik und Poliklinik), Hamburg
  - Universitätsklinikum Heidelberg (Medizinische Universitätsklinik/Innere Medizin IV/Nationales Centrum für Tumorerkrankungen), Heidelberg
  - Johannes Gutenberg-Universität Mainz (I. Medizinische Klinik und Poliklinik), Mainz
  - Klinikum rechts der Isar der Technischen Universität München (Medizinische Klinik und Poliklinik II/Gastroenterologie), Munich
  - Universitätsklinikum Tübingen (Medizinische Klinik/Innere Medizin I), Tübingen
- Italy (7):
  - l'Azienda Ospedaliero-Universitaria di Bologna-Policlinico S. Orsola Malpighi, Bologna
  - l'Università degli Studi di Genova (Dipartimento di Medicina Interna e Specialità Mediche), Genova
  - Istituto Europea di Oncologia EIO, Milan
  - A.O.R.N. Monaldi-Cotugno-CTO, Napoli
  - l'Azienda Ospedaliera di Padova and l'Istituto Oncologico Veneto IOV, Padua
  - l'Ente "Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone", Palermo
  - L'Istituto Clinico Humanitas-Humanitas Mirasole S.p.A., Rozzano-Milano

REFERENCES:
- [Derived] Bitzer M, Horger M, Giannini EG, Ganten TM, Worns MA, Siveke JT, Dollinger MM, Gerken G, Scheulen ME, Wege H, Zagonel V, Cillo U, Trevisani F, Santoro A, Montesarchio V, Malek NP, Holzapfel J, Herz T, Ammendola AS, Pegoraro S, Hauns B, Mais A, Lauer UM, Henning SW, Hentsch B. Resminostat plus sorafenib as second-line therapy of advanced hepatocellular carcinoma - The SHELTER study. J Hepatol. 2016 Aug;65(2):280-8. doi: 10.1016/j.jhep.2016.02.043. Epub 2016 Mar 4. PMID 26952006